CLINICAL TRIAL: NCT04172805
Title: A Single-arm, Open, Phase II Study of Anlotinib Combined With Toripalimab in Refractory and Advanced Soft-tissue Sarcoma
Brief Title: Anlotinib Combined With Toripalimab in Refractory and Advanced Soft-tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xing Zhang, Vice director of department of medical sarcoma and melanoma,Principal Investigator,Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SunYat-senU-anlotinib &pd-1
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Sarcoma,Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — anlotinib; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib combined with Toripalimab (Experimental): Anlotinib 12mg orally per day, two weeks on , one week off; 240 mg of toripalimab (fixed dose) every three weeks.
  Interventions: Drug: anlotinib and toripalimab

INTERVENTIONS:
Drug: anlotinib and toripalimab — Anlotinib 12mg orally per day, two weeks on , one week off; 240 mg of toripalimab (fixed dose) every three weeks. Repeat every three weeks. Patients with disease control (CR + PR + SD) and tolerable adverse reactions continued to take medication until the researchers concluded that patients were not suitable to continue medication or the efficacy evaluation was disease progression (PD). No other antineoplastic treatment can be given during the treatment.
  Other Names: Anlotinib Hydrochloride

SUMMARY:
Soft tissue sarcoma (STS) is a relatively rare type of malignant tumor with an incidence of 1-2/100000. For unresectable or widely disseminated advanced STS, a combined clinical trial is the best way to obtain evidence-based medical evidence.

Anlotinib, a multi-target receptor tyrosine kinase inhibitor (TKI), is effective for various histological types of STS and the safety is tolerable. TKIs may reverse drug resistance or inefficiency of immunoassay inhibitors, and combination therapy has shown preliminary efficacy in a variety of tumors.

Because of the poor prognosis of refractory and advanced STS, there is no standard second-line treatment. Therefore, combined therapies based on the original targeted drugs would be paid more concentrations in the future. We focus on exploring the feasibility of combination of anlotinib and Toripalimab monoclonal antibody in advanced, refractory and progressive soft tissue sarcoma after failure of standard treatment, and look forward to further improving the efficacy of soft tissue sarcoma.

DETAILED DESCRIPTION:
Soft tissue sarcoma (STS) is a relatively rare type of malignant tumor. For patients with recurrent/distant metastasis/unresectable advanced soft tissue sarcoma, chemotherapy with doxorubicin and ifosfamide is the standard treatment, but the effect is limited.

Targeted drugs represented by anti-angiogenesis targeted drugs have had certain clinical benefits in the treatment of sarcoma. Among them, anlotinib, a multi-target receptor tyrosine kinase inhibitor, is effective for STS of various tissue types and the safety is tolerable. Previous clinical studies have found that anlotinib has a certain effect on a variety of solid tumors including thyroid cancer, lung cancer, soft tissue sarcoma, and kidney cancer. In 2016, a phase II clinical study evaluated the efficacy and safety of anlotinib advanced STS, especially synovial sarcoma and alveolar soft tissue sarcoma. The study included 154 patients with evaluable efficacy, with an ORR of 10.13% and a median PFS of 5.63 months. Even so, the limited efficacy of targeted drugs remains a bottleneck. For advanced unresectable or widely disseminated soft tissue sarcomas, a combined clinical trial is the best way to obtain evidence-based medical evidence.

In recent years, anti-PD-1 antibodies have been reported as effective treatment in solid tumors, and their clinical application has become increasingly widespread. The anti-PD-1 antibody Toripalimab has also been listed recently, and its clinical application prospects are huge. Anti-PD-1 antibodies also have been proved effect better in combination with targeted therapies. Multiple in vitro studies have shown that low-dose anti-angiogenesis targeted drugs can reduce hypoxia, increase CD8+ T cell infiltration, reduce tumor-associated macrophage (TAM) recruitment in non-small cell lung cancer and reduce tumor and serum. The level of TGF-β is increased, thereby enhancing the anti-PD-1 antibody effect and significantly inhibiting tumor growth and metastasis. At the same time, by evaluating the therapeutic effects of combination therapy in other tumors, we aim to investigate that anti-angiogenesis targeted drugs combined with anti-PD-1 antibodies have considerable potential for sarcoma treatment.

At present, a number of clinical trials of anti-angiogenesis targeted drugs combined with anti-PD-1 antibody for tumor treatment are underway or will be carried out, but the clinical study of anti-PD-1 antibody with anlotinib has not yet started. In response to the above problems, the aim of this study was to explore the efficacy and to assess the safety of anti-PD-1 antibody in the treatment of refractory and advanced STS patients with first-line treatment failure, which would provide patients with STS better treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily joined the study and signed informed consent, with good adherence and follow-up.
2. Male or female patients aged 18-70 years, ECOG PS score: 0 to 2 points; expected survival over 3 months.
3. All advanced soft tissue sarcomas, first-line treatment failure or inability to tolerate first-line treatment, diagnosed by histology, at least one measurable lesion according to RECIST 1.1, including synovial sarcoma, leiomyosarcoma, alveolar soft tissue sarcoma, undifferentiated pleomorphic sarcoma/malignant fibrous histiocytoma, liposarcoma, fibrosarcoma, clear cell sarcoma, angiosarcoma, epithelioid sarcoma, malignant peripheral nerve sheath tumor, undifferentiated sarcoma, dermatofibrosarcoma, inflammatory myofibroblast sarcoma, malignant solitary fibroids. However, the following types can be treated first-line: alveolar soft tissue sarcoma, well differentiated / dedifferentiated / pleomorphic liposarcoma, clear cell sarcoma;
4. At least one target lesion measurable according to RECIST version 1.1 in the past 3 months, and in at least 1 direction (maximum diameter required to be recorded) can be obtained by magnetic resonance imaging (MRI) or computed tomography (CT) Accurate measurement, where conventional CT ≥ 20 mm or ≥ 10 mm under spiral CT.
5. The main organ function meets the following criteria within 7 days of treatment:

   * Blood routine examination criteria (without blood transfusion within 14 days): hemoglobin (HB) ≥ 90g / L; neutrophil absolute value (ANC) ≥ 1.5 × 109 / L; platelets (PLT) ≥ 80 × 109 / L.
   * Biochemical tests are subject to the following criteria: total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5ULN, such as with liver metastasis, then ALT and AST ≤ 5ULN; serum creatinine (Cr) ≤ 1.5ULN or creatinine clearance (CCr) ≥ 60ml / min;
   * Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low (50%).
6. Women of childbearing age must have taken reliable contraceptive measures and performed a pregnancy test (serum or urine) within 7 days prior to enrollment, and the results were negative, and were willing to use appropriate methods during the trial and 8 weeks after the last administration of the test drug. For men, consent must be given to the appropriate method of contraception or surgical sterilization during the trial and 8 weeks after the last administration of the test drug.

Exclusion Criteria:

1. Patients who have previously been treated with anlotinib or anti-PD-1/PD-L1 antibodies.
2. Exceeded or currently suffering from other malignant tumors within 5 years, with the exception of cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (in situ carcinoma) And T1 (tumor infiltrating basement membrane)].
3. Planning to use cytotoxic therapy, signal transduction inhibitors, immunotherapy (or mitomycin C used within 6 weeks prior to receiving the test drug) within 4 weeks prior to enrollment or during the study. Radiation-rehabilitation radiotherapy (EF-RT) was performed within 4 weeks prior to enrollment or limited-field radiotherapy to be evaluated for tumor lesions within 2 weeks prior to grouping.
4. Hair loss is not included due to unresolved toxicities above CTC AE Level 1 for any prior treatment.
5. A variety of factors that affect oral medications (such as inability to swallow, chronic diarrhea, and intestinal obstruction), and symptomatic treatment is uncontrollable.
6. With pleural effusion or ascites, causing respiratory syndrome (≥ CTC AE grade 2 dyspnea [level 2 dyspnea refers to short-term shortness of activity; affecting instrumental activities of daily living]), and symptomatic treatment is uncontrollable.
7. Active central nervous system (CNS) metastases with clinical signs including cerebral edema, steroid requirements, or progressive disease. Patients with previously treated brain or meningeal metastases must be clinically stable (magnetic resonance imaging [MRI] shows no evidence of new or enlarged metastases at least 4 weeks apart) and stop the immunosuppressant amount of systemic steroids (> 10 Mg / day) prednisone or equivalent) at least 2 weeks prior to study drug administration.
8. Patients with abnormal thyroid function after optimal drug treatment.
9. Patients with any severe and/or uncontrolled diseases, including:

   * Hypertension and uncontrollable levels of normal anti-hypertensive medication (within 3 months): systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg.
   * Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months prior to enrollment, unstable or severe angina, or coronary artery bypass surgery, congestive heart failure (New York Heart Association (NYHA) ) > 2), ventricular arrhythmia requires medical intervention, left ventricular ejection fraction (LVEF) <50%. Have grade I or higher myocardial ischemia or myocardial infarction, arrhythmia (including QTC ≥ 480ms) and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification);
   * Active or uncontrolled serious infection (≥ CTC AE Level 2 infection);
   * Objective evidence of previous or current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe impaired lung function, etc.
   * Liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral therapy;
   * Renal failure requires hemodialysis or peritoneal dialysis;
   * Patients with a history of any active autoimmune disease or autoimmune disease, including but not limited to the following: hepatitis, pneumonia, uveitis, colitis (inflammatory bowel disease), pituitary inflammation, vasculitis, nephritis, Hyperthyroidism and hypothyroidism, except for vitiligo patients to resolve or resolve childhood asthma / atopic disease. Asthma that requires intermittent use of bronchodilators or other medical interventions should also be excluded.
   * History of immunodeficiency includes human immunodeficiency virus (HIV) or other acquired or congenital immunodeficiency disease or active hepatitis (transaminase does not meet, hepatitis B virus (HBV) DNA ≥ 104/ml or hepatitis C virus) Seropositive (HCV) RNA ≥ 103/ml or higher); HBV DNA <2000 IU / ml (<104 / ml) carriers of chronic hepatitis B must receive antiviral therapy throughout the study period.
   * Need to use immunosuppressive drugs or immunosuppressive agents for systemic or concurrent medical conditions that can absorb local corticosteroids. Dosage > 10 mg / day prednisone or equivalent is prohibited within 2 weeks prior to study drug administration. Note: Corticosteroids for IV versus allergy prevention purposes are permitted.
   * Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L);
   * Urine routine indicates that urine protein ≥ ++, and confirmed 24-hour urine protein quantitation > 1.0 g;
   * Patients with seizures and need treatment;
   * abnormal blood coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolysis or anticoagulant therapy; Note: International standardization in prothrombin time Under the premise of an odds ratio (INR) ≤ 1.5, low-dose heparin (up to 0.6 million to 12,000 U per day for adults) or low-dose aspirin (daily dose ≤ 100 mg) is allowed for preventive purposes.
10. Major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to grouping.
11. Imaging studies show that the tumor has invaded the important perivascular circumference or that the patient is likely to invade the important blood vessels during the follow-up study and cause fatal bleeding.
12. Patients with any signs of hemorrhage or history, regardless of severity; patients with any bleeding or bleeding episodes ≥ CTCAE 3 within 4 weeks prior to grouping have unhealed wounds, ulcers, or fractures.
13. Overactive/venous thrombosis occurred within 6 months, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism.
14. Active infection or unexplained fever > 38.5 ° C during screening visits or on the first scheduled date of administration (subject to the subject's decision to recruit subjects with tumor fever).
15. Those who have a history of psychotropic substance abuse and are unable to quit or have a mental disorder.
16. Participated in other anti-tumor drug clinical trials within 4 weeks.
17. According to the investigator's judgment, there are people with concomitant diseases that seriously endanger the safety of the patient or affect the patient's completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Time Frame: each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Objective response rate is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.

SECONDARY OUTCOMES:
Progress free survival | Time Frame: until Progressive Disease (PD) or death (up to 24 months)
  Progress free survival is defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.
Overall Survival | Time Frame: From randomization until death (up to 24 months)
  Overall survival is defined as the time until death due to any cause.
Disease Control Rate | Time Frame: each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Xing Zhang, Guangzhou, Guangdong, China